CLINICAL TRIAL: NCT05627310
Title: Development and Validation of a Deep Learning System for Nasopharyngeal Carcinoma Using Endoscopic Images: a Multi-center Prospective Study
Brief Title: Development and Validation of a Deep Learning System for Nasopharyngeal Carcinoma Using Endoscopic Images
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Nanchang University (Other); Fujian Medical University Union Hospital (Other); Quan Zhou First Affiliated Hospital of Fujian Medical University (Unknown); First Affiliated Hospital of Guangxi Medical University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); The People' s Hospital of Jiangmen (Unknown)
Responsible Party: Sponsor
Other Study IDs: AIAD202204
Record Dates: First submitted 2022-07-11; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; deep learning; tumor screening
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training Cohort: Nasopharyngeal endoscopic images collected from 8 hospitals all over China
- Validation Cohort: Nasopharyngeal endoscopic images collected from 8 hospitals all over China
  Interventions: Other: Diagnostic
- Testing Cohort: Nasopharyngeal endoscopic images prospectively collected from 8 hospitals all over China
  Interventions: Other: Diagnostic

INTERVENTIONS:
Other: Diagnostic — Training dataset was used to train the deep learning model, which was validated and tested by external dataset.
  Groups: Testing Cohort; Validation Cohort

SUMMARY:
Develop a deep learning algorithm via nasal endoscopic images from eight NPC treatment centerto detect and screen nasopharyngeal carcinoma(NPC).

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is an epithelial cancer derived from nasopharyngeal mucosa. Nasal endoscopy is the conventional examination for NPC screening. It is a major challenge for inexperienced endoscopists to accurately distinguish NPC and other benign dieseases. In this study, we collcet multi-center endoscopic images and train a deep learning model to detect NPC and indicate tumor location. Then, the model perfomance will be compared with endoscopists and be tested prospectively with external dataset.

ELIGIBILITY:
Inclusion Criteria:

* The quality of endoscopic images should clinical acceptable.
* Patients were diagnosed with biopsy(NPC, benign hyperplasia). Control corhort(normal nasopharynx) don't require bispsy result.

Exclusion Criteria:

* images with spots from lens flares or stains, and overexposure were excluded from further analysis.
* image can not expose most part of lesion clearly.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nasopharyngeal endoscopic images were collected from 8 hospital in NPC epidemic area all over China.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve of the deep learning algorithm | baseline
  The investigators will calculate the area under the receiver operating characteristic curve of deep learning algorithm and compare this index between deep learning system and human doctors.

SECONDARY OUTCOMES:
Sensitivity of the deep learning system | baseline
  The investigators will calculate the sensitivity of deep learning algorithm and compare this index between deep learning system and human doctors.
Specificity of the deep learning system | baseline
  The investigators will calculate the specificity of deep learning algorithm and compare this index between deep learning system and human doctors.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, MD PhD, Principal Investigator — Eye&ENT Hospital, Fudan University
Locations (8):
- China (8):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Quan Zhou First Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The People' s Hospital of Jiangmen, Jiangmen, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The People' s Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Eye&ENT Hospital of Fudan University, Shanghai, Shanghai Municipality